CLINICAL TRIAL: NCT04927247
Title: A Randomized, Double-blind, Placebo-controlled, Multicenter Study of a Single Dose of Inclacumab to Reduce Re-admission in Participants With Sickle Cell Disease and Recurrent Vaso-occlusive Crises
Brief Title: A Study of a Single Dose of Inclacumab to Reduce Re-admission in Participants With Sickle Cell Disease and Recurrent Vaso-occlusive Crises
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study was terminated due to poor accrual and associated recrutiment challenges
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GBT2104-132; C5361002 (Other: Alias Study Number); 2020-005287-60 (EudraCT Number: CTIS (EU)); 2020-005287-60 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2021-05-26; First posted 2021-06-15 (Actual); Results first posted 2024-12-11 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-11

CONDITIONS: Sickle Cell Disease; Vaso-occlusive Crisis; Vaso-occlusive Pain Episode in Sickle Cell Disease
Keywords: Re-admission; Acute; blood disorders; hemoglobin; red blood cells; RBCs; sickle-like shape; mutation in hemoglobin gene; sickle-cell trait; sickle-cell crisis; Sickle Cell Disease; SCD; Vaso-occlusive Crisis; VOC; SCA
MeSH Terms: conditions — Anemia, Sickle Cell; Vaso-Occlusive Crises; Hematologic Diseases; Sickle Cell Trait | interventions — inclacumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double blind study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- inclacumab 30 mg/kg (Experimental): Inclacumab 30 mg/kg administered intravenously (IV)
  Interventions: Drug: Inclacumab
- placebo (Placebo Comparator): Placebo administered IV
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Inclacumab — Inclacumab will be supplied in single use 10 mL vials at a concentration of 50 mg/mL. One vial contains 500 mg of inclacumab. This is a liquid concentrate for IV infusion.
  Arms: inclacumab 30 mg/kg
Drug: Placebo — Placebo will be supplied in single use 10 mL vials containing the same ingredients without the active drug. Placebo will be prepared as a liquid concentrate for IV infusion and administered in the same manner as active study drug.
  Arms: placebo

SUMMARY:
This Phase 3 study will assess the safety and efficacy of a single dose of inclacumab, a P-selectin inhibitor, for a vaso-occlusive crisis (VOC) after an index VOC in participants with sickle cell disease (SCD). Participants will be randomized to receive either inclacumab or placebo.

DETAILED DESCRIPTION:
The study will include approximately 280 adult and adolescent participants (≥ 12 years of age) with SCD.

Eligible participants will be administered inclacumab or placebo intravenous (IV) as a single dose.

Participants that complete the study through Day 90 will be provided the opportunity to enroll in an open-label extension (OLE) study.

ELIGIBILITY:
Inclusion Criteria:

1. Participant has an index VOC. The index VOC is any VOC that required admission to a healthcare facility and treatment with parenteral pain medication. An admission for the index VOC includes:

   1. A hospital admission, or
   2. An admission to an emergency room, observation unit, or infusion center for ≥ 12 hours, or
   3. 2 visits to an emergency room, observation unit, or infusion center over a 72-hour period

   for an acute episode of pain with no other cause other than a vaso- occlusive event that includes the following:
   * Uncomplicated VOC,
   * Acute chest syndrome (ACS),
   * Acute hepatic sequestration,
   * Acute splenic sequestration, or
   * Priapism.
2. Participant has a confirmed diagnosis of SCD (any genotype). Documentation of SCD genotype is required and may be based on documented history of laboratory testing or confirmed by laboratory testing at Baseline.
3. Participant is male or female, ≥ 12 years of age at the time of informed consent.
4. Participant has experienced between 2 and 10 VOCs within the 12 months prior to Screening as determined by documented medical history. The index VOC is not to be considered as one of the 2 to 10 events. A prior VOC is defined as an acute episode of pain that:

   1. Has no medically determined cause other than a vaso-occlusive event, and
   2. Results in a visit to a healthcare facility (hospital, emergency department, urgent care center, outpatient clinic, or infusion center) or results in a remote contact with a healthcare provider; and
   3. Requires parenteral narcotic agents, parenteral nonsteroidal anti-inflammatory drugs (NSAIDs), or an increase in treatment with oral narcotics.
5. Participants receiving erythropoiesis-stimulating agents (ESA, e.g., erythropoietin [EPO]) must be on a stable dose for at least 90 days prior to Screening and expected to continue with the stabilized regimen throughout the course of the study.
6. Participants receiving hydroxyurea (HU), L-glutamine, or voxelotor (Oxbryta®) must be on a stable dose for at least 30 days prior to Screening and expected to continue with the stabilized regimen throughout the course of the study.

Exclusion Criteria:

1. Participant is receiving regularly scheduled red blood cell (RBC) transfusion therapy (also termed chronic, prophylactic, or preventative transfusion).
2. Participant is taking or has received crizanlizumab (ADAKVEO®) within 90 days prior to Screening.
3. Participant weighs > 133 kg (292 lbs.).

Other protocol-defined Inclusion/Exclusion may apply.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2021-12-09 (Actual); Primary Completion 2023-11-24 (Actual); Study Completion 2023-11-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (59):
- United States (17):
  - Strada Patient Care Center, Mobile, Alabama
  - University of South Alabama Children's and Women's Hospital, Mobile, Alabama
  - University of South Alabama Mitchell Cancer Institute, Mobile, Alabama
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - UCSF Benioff Children's Hospital, Oakland, Oakland, California
  - Children's Hospital of Orange County, Orange, California
  - St. Joseph's Hospital, Tampa, Florida
  - University of Michigan Hospitals - Michigan Medicine, Ann Arbor, Michigan
  - Functional Fluidics, Inc., Detroit, Michigan
  - Alliance for Childhood Diseases dba Cure 4 The Kids Foundation, Las Vegas, Nevada
  - Erie County Medical Center, Buffalo, New York
  - Jacobi Medical Center, The Bronx, New York
  - Duke University Medical Center, Durham, North Carolina
  - DUMC Investigational Drug Services Pharmacy, Durham, North Carolina
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - PPD Bioanalytical, Richmond, Virginia
- Brazil (8):
  - Instituto D'Or de Pesquisa e Ensino - Hospital São Rafael, Salvador, Estado de Bahia
  - Multihemo Servicos Medicos S/A, Recife, Pernambuco
  - Hospital de Clinicas de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Fundação Faculdade Regional de Medicina de São José do Rio Preto, São José do Rio Preto, São Paulo
  - Casa de Saude Santa Marcelina, São Paulo, São Paulo
  - Instituto Estadual de Hematologia Arthur de Siqueira Cavalcanti - HEMORIO, Rio de Janeiro
  - Hospital das Clínicas da Faculdade de Medicina da Universidade de São Paulo -HCFMUSP, São Paulo
  - CEPEC-Centro de Pesquisa Clinica, São Paulo
- Colombia (2):
  - Clinica de la Costa Ltda., Barranquilla, Atlántico
  - Organizacion Clinica Bonnadona Prevenir S.A.S., Barranquilla, Atlántico
- France (2):
  - Hopital Avicenne, Bobigny
  - Hopital Henri Mondor, Créteil
- Universitatsklinikum Regensburg Padiatrische Hamatologie, Onkologie und Stammzelltransplantation, Regensburg, Germany
- Italy (6):
  - Farmacia Interna Azienda Ospedaliero-Ente Ospedaliero Ospedali Galliera, Genova, Genoa
  - S.S.D. Microcitemia, anemie congenite e dismetabolismo del ferro, Genova
  - DAI Materno-Infantile, UOC Clinica Pediatrica 1 Azienda Ospedaliera Universitaria "Luigi Vanvitell, Napoli
  - UO di Farmacia Clinica, Dipartimento di Medicina Sperimentale Azienda Ospedaliera Universitaria, Napoli
  - UOC Patologia Clinica e Molecolare Azienda Ospedaliera Universitaria "Luigi Vanvitelli", Napoli
  - UOC Radiologia Azienda Ospedaliera Universitaria "Luigi Vanvitelli", Napoli
- Kenya (4):
  - Kemri/Crdr, Siaya, Kemri Clinical Research Annex,, Kisumu, Siaya County
  - International Cancer Institute, Eldoret
  - Kenya medical Research Institute-centre for Respiratory Disease Research, Nairobi
  - Strathmore University Medical Center - Center for Research in Therapeutic Sciences(CREATES), Nairobi
- Lebanon (2):
  - American University of Beirut Medical Center, Hamra, Beyrouth
  - Nini Hospital, Tripoli, North Lebanon
- Nigeria (8):
  - University of Calabar Teaching Hospital, Calabar, Cross River State
  - National Hospital Abuja, Abuja, Federal Capital Territory
  - University of Abuja Teaching Hospital, Gwagwalada, Federal Capital Territory
  - Ahmadu Bello University Teaching Hospital (ABUTH), Zaria, Kaduna State
  - University of Nigeria Teaching Hospital, Enugu
  - Barau Dikko Teaching Hospital/Kaduna State University, Kaduna
  - Aminu Kano Teaching Hospital, Kano
  - Department of Pediatrics, College of Medicine, Lagos University Teaching Hospital, Lagos
- Sultan Qaboos University Hospital, Muscat, Oman
- Prince Mohammed bin Nasser Hospital, Jizan, Southern, Saudi Arabia
- Turkey (Türkiye) (4):
  - Hacettepe University, Ankara, Altindag/sihhiye
  - Mersin Universitesi Tip Fakultesi Saglik Arastirma ve Uygulama Merkezi Hastanesi, Yenischir, Mersin, Mersin
  - Baskent University Hospital, Adana, Yuregir
  - Acibadem Adana Hastanesi Cocuk Hematoloji Onkoloji, Adana
- Guy's & Thomas' NHS Foundation Trust, London, England, United Kingdom
- Zambia (2):
  - Matero Clinical Research Site,, Lusaka
  - University Teaching Hospital- Children's Hospital, Lusaka

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=GBT2104-132

RESULTS

PARTICIPANT FLOW:
Recruitment Details: In this study, participants with sickle cell disease (SCD), aged greater than or equal to (>=) 12 years were randomized to receive either inclacumab or placebo for reducing the frequency of re-admissions due to vaso-occlusive crisis (VOC) after an index VOC.
Pre-assignment Details: A total of 72 participants were enrolled and randomized in the study.
Groups:
- Inclacumab 30 mg/kg: Participants were administered with inclacumab 30 milligram per kilogram (mg/kg) intravenous (IV) infusion on Day 1 as a single dose.
- Placebo: Participants were administered with placebo IV infusion on Day 1 as a single dose.
Period: Overall Study
Arm/Group | Inclacumab 30 mg/kg | Placebo
Started | 37 | 35
Completed | 34 | 33
Not Completed | 3 | 2
Not completed — Other | 2 | 1
Not completed — Physician Decision | 0 | 1
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Population: The intent-to-treat (ITT) population included all randomized participants.
Groups:
- Inclacumab 30 mg/kg: Participants were administered with inclacumab 30 mg/kg IV infusion on Day 1 as a single dose.
- Total: Total of all reporting groups
Arm/Group | Inclacumab 30 mg/kg | Placebo | Total
Number analyzed (Participants) | 37 | 35 | 72
Age, Continuous [Mean (Standard Deviation); unit: Years] | 23.5 (6.95) | 24.9 (8.34) | 24.2 (7.64)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 17 | 39
  Male | 15 | 18 | 33
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 2 | 5
  Not Hispanic or Latino | 33 | 33 | 66
  Unknown or Not Reported | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With at Least 1 VOC That Required Admission to a Healthcare Facility and Treatment With Parenteral Pain Medication Within 90 Days of Randomization
Description: A VOC was a complication of SCD characterized by vaso-occlusion presenting as recurrent pain episodes. An admission for a VOC included a hospital admission, or an admission to an emergency room, observation unit, or infusion center for >= 12 hours, or 2 visits to an emergency room, observation unit, or infusion center over a 72-hour period. An acute episode of pain with no other cause other than a vaso-occlusive event included: uncomplicated VOC, acute chest syndrome, hepatic sequestration, splenic sequestration, or priapism. All on-study VOCs were adjudicated by an independent, blinded VOC Adjudication Committee comprised of experts in SCD.
Time Frame: Within 90 days of randomization (randomization happened on Day 1 [Day 1 to Day 91])
Population: The intent-to-treat (ITT) population included all randomized participants. Participants without an observed VOC who discontinued the study prior to Day 91 were assumed to have experienced at least one VOC.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Inclacumab 30 mg/kg | Placebo
Number analyzed (Participants) | 37 | 35
Percentage of participants | 45.4 (28.7) [28.7 to 62.2] | 37.5 (20.7) [20.7 to 54.3]
Statistical Analysis 1: Comparison: Inclacumab 30 mg/kg vs Placebo; Test type: Other; p = 0.6302, Exact Cochran-Mantel-Haenszel test; Difference in percentage = 7.9, 95% CI 2-sided [-15.8 to 31.7]

2. Secondary Outcome: Time to First VOC That Required Admission to a Healthcare Facility and Treatment With Parenteral Pain Medication Within 90 Days of Randomization
Description: A VOC was a complication of SCD characterized by vaso-occlusion presenting as recurrent pain episodes. Time to first VOC that required admission to a healthcare facility and treatment with parenteral pain medication within 90 days was defined as the time between randomization date and onset date of first VOC event. For participants who did not experience a protocol-defined VOC within 90 days of randomization, time to first VOC was censored at the end of their time at risk (participant's end of study date or Study Day 91, whichever was earlier). An admission for a VOC included a hospital admission, or an admission to an emergency room, observation unit, or infusion center for >= 12 hours, or 2 visits to an emergency room, observation unit, or infusion center over a 72-hour period. All on-study VOCs were adjudicated by an independent, blinded VOC Adjudication Committee comprised of experts in SCD. Kaplan-Meier method used for analysis.
Time Frame: Within 90 days of randomization (randomization happened on Day 1 [Day 1 to Day 91]) or censored day, whichever occurred earlier
Population: The ITT population included all randomized participants.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Inclacumab 30 mg/kg | Placebo
Number analyzed (Participants) | 37 | 35
Days | NA [NA to NA] — Here "NA" indicates that data could not be estimated as the number of participants with events available was not sufficient for the calculation of median and 95% CI using Kaplan-Meier method. | NA [NA to NA] — Here "NA" indicates that data could not be estimated as the number of participants with events available was not sufficient for the calculation of median and 95% CI using Kaplan-Meier method.
Statistical Analysis 1: Comparison: Inclacumab 30 mg/kg vs Placebo; Test type: Other; p = 0.9382, Stratified log-rank test; Hazard Ratio (HR) = 0.97, 95% CI 2-sided [0.43 to 2.16]

3. Secondary Outcome: Percentage of Participants With at Least 1 VOC That Required Admission to a Healthcare Facility and Treatment With Parenteral Pain Medication Within 30 Days of Randomization
Description: as for outcome 1
Time Frame: Within 30 days of randomization (randomization happened on Day 1 [Day 1 to Day 31])
Population: The ITT population included all randomized participants. Participants without an observed VOC who discontinued the study prior to Day 31 were assumed to have experienced at least one VOC.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Inclacumab 30 mg/kg | Placebo
Number analyzed (Participants) | 37 | 35
Percentage of participants | 8.2 (0.0) [0.0 to 17.3] | 25.0 (9.6) [9.6 to 40.4]
Statistical Analysis 1: Comparison: Inclacumab 30 mg/kg vs Placebo; Test type: Other; p = 0.1143, Exact Cochran-Mantel-Haenszel test; Difference in percentage = -16.8, 95% CI 2-sided [-34.4 to 0.8]

4. Secondary Outcome: Rate of VOCs Leading to a Healthcare Visit That Requires Parenteral Pain Medication or an Increase in Treatment With Oral Narcotics Within 90 Days Following Randomization
Description: VOC leading to a healthcare visit was defined as VOC at (hospital, emergency room, clinic visit, or remote contact with a healthcare provider) that required parenteral pain medication (e.g., parenteral narcotic agents or parenteral nonsteroidal anti-inflammatory drugs [NSAIDs]), or an increased treatment with oral narcotics. Complicated VOCs included acute chest syndrome (ACS),hepatic sequestration, splenic sequestration, and priapism. For each participant, the time period at risk for evaluation of VOCs was from date of randomization to the participant's end of study date or study Day 91, whichever was earlier. In this outcome measure adjusted rates of VOCs (percentages) reported were based on estimate from a negative binomial model with the independent variable of treatment group (inclacumab, placebo) and adjusted for baseline hydroxyurea use (yes, no). All on-study VOCs were adjudicated by an independent, blinded VOC Adjudication Committee comprised of experts in SCD.
Time Frame: Within 90 days of randomization (randomization happened on Day 1 [Day 1 to Day 91])
Population: The ITT population included all randomized participants.
Measure: Number (95% Confidence Interval); unit: Percentage of VOCs
Arm/Group | Inclacumab 30 mg/kg | Placebo
Number analyzed (Participants) | 37 | 35
Percentage of VOCs | 0.83 (0.57) [0.57 to 1.21] | 0.76 (0.51) [0.51 to 1.14]
Statistical Analysis 1: Comparison: Inclacumab 30 mg/kg vs Placebo; Test type: Other; p = 0.7549, Negative binomial model; Rate ratio = 1.09, 95% CI 2-sided [0.63 to 1.89]

ADVERSE EVENTS:
Time Frame: Day 1 through Day 161
Description: Safety population included randomized participants who received treatment with study drug.
Arm/Group | Inclacumab 30 mg/kg | Placebo
All-Cause Mortality (participants affected / at risk) | 1/36 | 0/33
Serious Adverse Events (participants affected / at risk) | 4/36 | 1/33
Other Adverse Events (participants affected / at risk) | 20/36 | 11/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Inclacumab 30 mg/kg (N=36) | Placebo (N=33)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Malaria (Infections and infestations) | 1 (1) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Inclacumab 30 mg/kg (N=36) | Placebo (N=33)
Sickle cell anaemia with crisis (Blood and lymphatic system disorders) | 2 (3) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Splenomegaly (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 1 (2) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Conjunctivitis allergic (Eye disorders) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Odynophagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0)
Hypothermia (General disorders) | 1 (1) | 0 (0)
Malaise (General disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0)
Peripheral swelling (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 1 (1)
Hypertransaminasaemia (Hepatobiliary disorders) | 2 (2) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 (1) | 0 (0)
Malaria (Infections and infestations) | 5 (6) | 3 (3)
Upper respiratory tract infection (Infections and infestations) | 2 (3) | 2 (2)
Urinary tract infection (Infections and infestations) | 2 (2) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Conjunctivitis (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Oral candidiasis (Infections and infestations) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Rhinovirus infection (Infections and infestations) | 1 (1) | 0 (0)
Sexually transmitted disease (Infections and infestations) | 1 (1) | 0 (0)
Acarodermatitis (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (3) | 1 (2)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (3)
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 4 (5) | 1 (1)
Dizziness (Nervous system disorders) | 2 (2) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Menstruation irregular (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publication until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2021-03-08): https://cdn.clinicaltrials.gov/large-docs/47/NCT04927247/Prot_000.pdf
  • Statistical Analysis Plan (2023-08-10): https://cdn.clinicaltrials.gov/large-docs/47/NCT04927247/SAP_001.pdf